CLINICAL TRIAL: NCT01043601
Title: A Phase IIb, Multi-center, Randomized, Double-blind, Placebo-controlled, Multi-dose, Four-period, Cross-over Study of Two Doses of Formoterol Fumarate MDI (PT005; 7.2 and 9.6 µg Ex-actuator), Administered Twice Daily for 1 Week in Patients With Moderate to Very Severe COPD, Compared to Open Label Marketed Formoterol Fumarate Inhalation Powder (Foradil® Aerolizer®, 12 µg) as an Active Control
Brief Title: Efficacy and Safety of Two Doses of Formoterol Fumarate MDI (PT005) in Patients With Stable Chronic Obstructive Pulmonary Disease (COPD), Compared to Foradil® Aerolizer® as an Active Control
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Similar data obtained in another study [see NCT01085045], therefore study not implemented.
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Chief Medical Officer, Pearl Therapeutics, Inc.
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PT0051002
Record Dates: First submitted 2010-01-05; First posted 2010-01-07 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Inhaled PT005 7.2 µg (Experimental)
  Interventions: Drug: Inhaled PT005
- Inhaled PT005 9.6 µg (Experimental)
  Interventions: Drug: Inhaled PT005
- Inhaled Placebo (Placebo Comparator)
  Interventions: Drug: Inhaled Placebo
- Formoterol Fumarate 12 µg (Foradil Aerolizer) (Active Comparator)
  Interventions: Drug: Formoterol Fumarate 12 µg (Foradil Aerolizer)

INTERVENTIONS:
Drug: Inhaled PT005 — inhaled, twice daily for 1 week duration
  Arms: Inhaled PT005 7.2 µg; Inhaled PT005 9.6 µg
Drug: Inhaled Placebo — inhaled, twice daily for 1 week duration
  Arms: Inhaled Placebo
Drug: Formoterol Fumarate 12 µg (Foradil Aerolizer) — inhaled, twice daily for 1 week duration
  Arms: Formoterol Fumarate 12 µg (Foradil Aerolizer)

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of inhaled formoterol fumarate (7.2 and 9.6 µg ex-actuator) compared to placebo and Foradil Aerolizer in patients with moderate to very severe chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Key Inclusion Criteria:

* Signed written informed consent
* 40 - 80 years of age
* Fluency in written and spoken English
* Females of non-child bearing potential or females of child bearing potential with negative pregnancy test; and acceptable contraceptive methods
* Current/former smokers with at least a 10 pack-year history of cigarette smoking
* A measured post- bronchodilator FEV1/FVC ratio of < or = 0.70
* A measured post- bronchodilator FEV1 > or = 750ml or 30% predicted and < or = 80% of predicted normal values
* Competent at using the inhalation device

Key Exclusion Criteria:

* Women who are pregnant or lactating
* Primary diagnosis of asthma
* Alpha-1 antitrypsin deficiency as the cause of COPD
* Active pulmonary diseases
* Prior lung volume reduction surgery
* Abnormal chest X-ray (or CT scan) not due to the presence of COPD
* Hospitalized due to poorly controlled COPD within 12 weeks of Screening
* Poorly controlled COPD, defined as the occurrence of acute worsening of COPD requiring corticosteroids or antibiotics or acute worsening of COPD requiring treatment prescribed by a physician within 6 weeks of screening or between screening and visit 2
* Lower respiratory tract infection requiring antibiotics within 6 weeks of screening
* Clinically significant medical conditions that preclude participation in the study (e.g. clinically significant abnormal ECG or uncontrolled hypertension)
* Positive Hepatitis B surface antigen or Hepatitis C antibody
* Cancer that has not been in complete remission for at least 5 years
* History of hypersensitivity to any beta2-agonists or any study drug component
* History of severe milk protein allergy
* Known or suspected history of alcohol or drug abuse
* Medically unable to withhold short acting bronchodilators for 8-hours
* Use of prohibited medications prior to screening and during the study as specified in the protocol
* Receiving long-term-oxygen or nocturnal oxygen therapy for >12 hours a day
* Participation in acute phase of pulmonary rehabilitation within 4 weeks of screening or will enter acute phase of pulmonary rehabilitation program during study
* Unable to comply with study procedures
* Prior participation in a Pearl PT005 study
* Requires use of a spacer due to poor hand-to-breath coordination

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-07; Primary Completion 2011-04 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Change in forced expiratory volume in one second (FEV1) area under the curve from 0 to 12 hours [AUC(0-12)] from test day baseline across the two doses of inhaled PT005 compared with placebo. | Day 7

SECONDARY OUTCOMES:
Lung Function Measures on Day 7 as measured by spirometry. | Day 7
Safety measures including electrocardiograms (ECGs), vital signs, physical exam, clinical laboratory testing, and adverse events of special interest | Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Charles Fogarty, MD, Principal Investigator — Spartanburg Medical Research
Locations (1):
- Spartanburg Medical Research, Spartanburg, South Carolina, United States